CLINICAL TRIAL: NCT06318949
Title: Albumin Modifications as Early Biomarkers of Chronic Liver Diseases
Acronym: MALAHBAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI22_0007 (MALAHBAR)
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Liver Disease
Keywords: predictive early biomarkers; albumine modifications; liver damage
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective multicentre study of biomarker validation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental)
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — If the patient does not object to participating in the study, a blood sample is taken at each visit (an additional tube may be added to a routine blood sample taken for standard care), or a residual blood sample is reused after routine tests have been performed, and data is collected from the medical record.

SUMMARY:
Chronic liver diseases, affecting over 800 million people worldwide, lead to approximately 2 million annual deaths. The need for early, sensitive diagnostic strategies to prevent disease progression and reduce mortality is still unmet. The traditional serum markers lack sensitivity and specificity, leading to the integration of these biomarkers into panel tests with algorithms or imaging measures. Despite their widespread use, these tests have limitations at an individual level, including an inability to predict disease progression or response to treatment. To address these shortcomings, our project proposes utilizing albumin post-translational modifications (PTM) as a predictive biomarker for liver disease progression. The hypothesis is that albumin modifications occur in the early stages of hepatocellular damage and are indicative of future liver diseases. These modifications can be detected through serum albumin isoform determination, albumin isoforms profiles or the albumin's ligand-binding capacities. Innovatively, the study will use the Serum Enhanced Binding (SEB) test, which identifies reduced ligand-binding capacities, and discusses a second patent for determining a typical isoform profile based on the hepatic injury type.

Our preliminary results from animal models and a proof-of-concept studies with patients support this hypotheses. Our previous studies demonstrated also significant differences in albumin isoform profiles in response to different types of hepatic injury and high sensitivity and specificity in the SEB test among cirrhotic patients.

The primary objective of the MALAHBAR project is to evaluate the capacity of albumin PTM to predict liver disease progression over three years in chronic liver disease patients. Secondary objectives include assessing the predictive ability of different albumin isoforms and the SEB test for liver disease progression, evaluating diagnostic performances and confirming characteristic albumin isoform profiles related to specific hepatic injuries. The study could represent a significant advancement in liver disease diagnostics and management, offering new insights into the role of albumin in liver pathology.

DETAILED DESCRIPTION:
More than 800 million people suffer from chronic liver disease (CLD) with approximately 2 million deaths per year. The progression of CLD, could be asymptomatic until the appearance of fibrosis, cirrhosis and sometimes hepatocellular carcinoma. The prevention and early diagnosis of liver disease is therefore a major public health issue.

Due to their lack of sensitivity and specificity, direct serum markers are now combined in " panel tests ", sometimes gathered and used in algorithms (FibroMeter, FibroTest, FIBROSpect, Hepascore…) to help diagnose fibrosis or cirrhosis and to assess the stage of liver damage. Other biomarkers, in particular molecules involved in the fibrosis process, (protein-based biomarkers, microRNA or collagen-based biomarkers) have been the subject of numerous studies, but have not yet led to clinically exploitable biomarkers for the medium- or long-term monitoring of CLD. Non-invasive, sensitive and specific biomarkers for the early detection of liver dysfunction leading to advanced liver disease are therefore still awaited.

It has been shown that chemical and structural modifications of human serum albumin (HAS) leading to different isoforms could be used as biomarkers for advanced liver disease. Our work supports the hypothesis that the main changes in HSA occur in the early stages of cellular liver damage and could be predictive of future liver disease. These modifications can be revealed by the profile of isoforms in the patient's serum, or even more efficiently by the binding capacities of HAS for different ligands with specific binding sites. On this basis, a patent application has been filed for the SEB (Serum enhanced binding) test.

The study plans to recruit 756 patients in 6 university hospital centers (CHU of Limoges, Angers, Poitiers, Tours, Rennes, and Pointe à Pitre). The recruitment period is of 1.5 year.

Each patient will be followed during 3 years maximumThe study requires no supplementary visit as compared to the standard care. Study visits will take place during usual visits of the standard care as follows:.

* Inclusion visit : study information by the investigator and if the patient is not opposed to participate to the study, either blood sampling (a supplementary tube can be add to a routine blood sampling realised for standard cares) or re-use of a residual blood sample after routine tests have been done, and data collection from the medical file.
* Follow-up visits: visits at 1, 2 and 3 years depending to the diagnostic of the investigator. During these visits: collection of a blood sampling the same conditions described for the inclusion visit and data collection from the medical file.

The samples will be sent to the central laboratory in the CHU of Limoges (Pharmacology, Toxicology and Pharmacovigilance) where HSA isoforms will be analysed by LC-QTOF and SEB tests realised.

The main goal is to validate HAS modifications as biomarker able to predict the evolution of liver damage and thus prevent worsening of the liver disease and finally improve the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* With a compensated fibrosis defined by an hepatic elasticity ≥10 kPa measured by FibroScan®
* Having had blood test at the hospital as part of a consultation or an hospitalisation at the inclusion including usual parameters for the liver disease follow-up
* Affiliated with or beneficiaries of a social security system
* Not opposed to participate to the study after being informed

Exclusion Criteria:

* Patients suffering from decompensated cirrhosis or with an history of decompensated cirrhosis
* Patients who received an albumin infusion in the month before the inclusion visit
* Patients suffering from stage 4 or 5 renal failure (GFR < 29 ml/min/1,73m²)
* Patients suffering from cancer
* Pregnant or breastfeeding women or women of childbearing age without effective contraception (based on declaration)
* Patients suffering from impairment of mental faculties or a psychiatric disorder which could interfere with the understanding of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Ability of HSA PTM to predict the evolution of liver damage at 3 year in patients with an advanced chronic liver disease (ACLD) as recently defined in the BAVENO VII recommendations based on FibroScan. | Years 3
  The primary outcome is the positive predictive value (VPP) of post-translational HSA modifications related to the worsening of the liver damage at 3 years . This will be determined by an augmentation of more than 20% as compared to the initial state, documented by FibroScan® or a liver related event as defined in BAVENO VII.

SECONDARY OUTCOMES:
ability of post-translational HSA modifications to predict the evolution of liver damage at 3 years based on liver-related events or on the worsening of the disease stage evaluated by the de Child Pugh or MELD score. | Year 3
  Positive predictive value (VPP) of post-translational HSA modifications related to the worsening of the liver damage at 3 years. This will be determined by the occurrence of one or several events of the following:
  1. Liver-related events
  2. Worsening of the disease stage evaluated by the Child Pugh score or of 2 points of the MELD score in case of cirrhosis.
ability of the different isoforms of HSA to predict the evolution of liver damage at 1 and 2 years provided that data are available in the medical file. | year 2
  Positive predictive value (VPP) of post-translational HSA modifications related to the worsening of the liver damage at 1 and 2 years. This will be determined by the occurrence of one or several events of the following
ability of SEB test to predict the evolution of liver damage at 3 years (and at 1 and 2 years provided data are available in the medical file). | Year 3
  Positive predictive value of the SEB test related to the worsening of the liver damage at 3 years, and at 1 and 2 years provided data are available in medical files.
diagnostic performances of the SEB test and of the different isoforms of HSA at each stage of the liver disease. | year 3
  Sensibility and specificity of the SEB test and of the different isoforms of HAS, at each stage of the . liver disease (Child Pugh A5, A6, B7, B8, B9, et > C10).
confirm that the isoforms of HAS present in the characteristic patterns (type of isoform and intensity) of the nature of the liver damage. | Years 3
  Ability to discriminate patients depending on the cause of the initial liver damage, taking into account the whole patterns of isoforms (including minor isoforms), with calculation of sensibility and specificity.

CONTACTS AND LOCATIONS:
Locations (7):
- France (6):
  - Angers Univeristy Hospital, Angers
  - Limoges University Hospital, Limoges
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours
- Pointe à Pitre University Hospital, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No